CLINICAL TRIAL: NCT06890468
Title: Three-in-One Stop Computed Topography Angiography and CT Perfusion in Cerebrovascular Disease
Brief Title: Three-in-One Stop Computed Topography Angiography(CTA) and CT Perfusion(CTP) in Cerebrovascular Disease
Status: Not yet recruiting | Type: Observational
Sponsor: Xin Lou (Other)
Responsible Party: Sponsor-Investigator, Xin Lou, Chairman, Chinese PLA General Hospital
Organization: Chinese PLA General Hospital (Other)
Other Study IDs: 301-CTAP
Record Dates: First submitted 2025-03-15; First posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Radiology; Vascular Diseases
Keywords: CTP; head and neck CTA
MeSH Terms: conditions — Vascular Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This research takes patients with cerebrovascular diseases as the research subjects and employs the experimental design of a prospective cohort study, aiming to innovatively develop and validate a "one-stop" multimodal CT examination scheme. The 301-CTAP multimodal CT technique implies that three modalities are acquired through a single collection, including head and neck CTA (head and neck CTA), multiphase CTA imaging of the brain (multiphase CTA), and CT perfusion imaging of the brain (CT perfusion).

DETAILED DESCRIPTION:
In the diagnosis of cerebrovascular diseases, CT examination, with its advantages of high resolution, non-invasiveness, and rapid imaging, has long become an indispensable diagnostic tool. Especially in the "Chinese Guidelines for the Standardized Application of Cerebrovascular Disease Imaging", the "one-stop" CT examination mode - including CT plain scan (NCCT), CT angiography (CTA), and CT perfusion imaging (CTP) - has been strongly recommended as the preferred imaging examination method for suspected acute large artery occlusion ischemic cerebrovascular diseases. However, traditional multimodal CT examinations require large amounts of contrast agents, multiple scans for blood flow and vascular imaging, multiple injections of contrast agents, high radiation doses, and low image signal-to-noise ratios. How to simultaneously evaluate cerebral blood flow perfusion and cerebral vessels through a single examination is a major clinical need that urgently needs to be addressed.

This study takes patients with cerebrovascular diseases as the research subjects and adopts a prospective cohort study design. The aim is to innovatively develop and verify a "one-stop" multimodal CT examination scheme. The 301-CTAP multimodal CT technology means that the three modalities are obtained through a single acquisition, including head and neck CTA (CTA), multiphase CTA (CTA) imaging of the brain, and CT perfusion imaging of the brain. The 301-CTAP multimodal CT technology can reduce the duration of CT examination for patients with cerebrovascular diseases without reducing the imaging content, and reduce the amount of contrast agents, X-ray radiation dose, and the incidence of contrast agent allergy and related adverse events. It provides innovative and important technical support for the diagnosis and assessment of acute stroke and other cerebrovascular emergencies; the acquisition of multiple key imaging indicators features enables individualized comprehensive imaging assessment, prediction of clinical functional prognosis and stroke recurrence risk for patients; the implementation of this project helps optimize the imaging examination path in the diagnosis and treatment of cerebrovascular diseases.

ELIGIBILITY:
Inclusion Criteria:

* Age≥18 <100years
* Head and neck artery stenosis/occlusion, moyamoya disease, aneurysm, artery dissection, etc., may include patients with acute stroke, chronic cerebral ischemia, and asymptomatic patients. After clinical assessment, CT perfusion imaging is required
* The image quality meets the requirements of diagnosis and post-processing
* Patients who follow the scanning strategy to complete the examination
* The patient or his or her family agrees to provide clinical data and follow-up
* Patients or their families sign informed consent forms

Exclusion Criteria:

* < 18 years old
* People who are allergic to iodine contrast agents, or who cannot be tested temporarily due to taking metformin or aminoglycoside drugs
* Renal failure patient
* Severe cardiac insufficiency
* Severe liver damage
* Patients with an expected survival of less than 1 year
* Patients with cerebrovascular diseasePregnant woman

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with cerebrovascular disease
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-03-16 (Estimated); Primary Completion 2029-12-30 (Estimated); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
Three-in-One Stop Computed Topography Angiography and Perfusion（301-CTAP） in the diagnosis of cerebrovascular disease performance description | 2 years
  Three-in-One Stop computed topography angiography and computed topography perfusion in cerebrovascular disease performance, including lesions in the detection and imaging in the diagnosis of image quality, accuracy, sensitivity and specificity.

CONTACTS AND LOCATIONS:
Overall Officials: Xin Lou, Study Chair — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing 100853, Beijing, China